CLINICAL TRIAL: NCT02666508
Title: A Randomized Trial of Plaque Identifying Toothpaste on Reduction of Plaque and Inflammation
Brief Title: Trial of Toothpaste to Reduce Plaque and Inflammation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Illinois at Chicago (Other)
Collaborators: Florida Atlantic University (Other)
Responsible Party: Principal Investigator, Kim Fasula, Director of Clinic Operations & Clinical Instructor, College of Dentistry, University of Illinois at Chicago
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2015-0620
Record Dates: First submitted 2016-01-24; First posted 2016-01-28 (Estimated); Results first posted 2021-01-14 (Actual); Last update posted 2021-01-14 (Actual); Status verified 2021-01

CONDITIONS: Plaque; Inflammation
Keywords: plaque identifying toothpaste; plaque score; C-reactive protein
MeSH Terms: conditions — Plaque, Amyloid; Inflammation

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- Plaque identifying toothpaste (Active Comparator): A 30 day supply of daily syringes containing a plaque identifying toothpaste with targetol
  Interventions: Other: Plaque identifying toothpaste
- Non-plaque identifying toothpaste (Active Comparator): A 30 day supply of daily syringes containing an identical non plaque identifying toothpaste without targetol
  Interventions: Other: Non-plaque identifying toothpaste

INTERVENTIONS:
Other: Plaque identifying toothpaste — Plaque identifying toothpaste with targetol
  Arms: Plaque identifying toothpaste
Other: Non-plaque identifying toothpaste — Non-plaque identifying toothpaste without targetol
  Arms: Non-plaque identifying toothpaste

SUMMARY:
Dental plaque causes caries and periodontal disease and data are sparse about toothpaste and plaque removal. Inflammation, caused by dental plaque, is a risk factor for cardiovascular disease. (CVD) The availability of (Plaque HD (TM), a plaque identifying toothpaste with targetol technology (TM)), afforded the unique opportunity to test whether there were statistically significant and clinically important reductions in plaque and inflammation in a randomized trial of apparently healthy individuals.

DETAILED DESCRIPTION:
The protocol was approved by the Institutional Review Board of the University of Illinois and the trial was posted on ClinicalTrials.gov. We screened all potentially eligible subjects from the Medical District of the University of Illinois which includes the Colleges of Dentistry, Medicine, Public Health and Pharmacy.

All willing and eligible subjects signed informed consent forms and were instructed to refrain from brushing or flossing teeth, using any oral hygiene aids (such as mouthwash or chewing gum) the evening prior to and the morning of the data collection appointment. All subjects were be asked to complete the following procedures:

1. Rinse for 10 seconds with 25 mL of phosphate buffer
2. Rinse for 1 minute with 5.0 mL of 1240-ppm fluorescein in phosphate buffer
3. Rinse 3 times (for 10 seconds) with 25mL of phosphate buffer
4. Be positioned on a tripod chin rest 15 inches in front of the camera, retraction placed and intraoral images captured under UV LED light imaging.
5. Provide a blood sample for hs-CRP.
6. Use a 30 day supply of their assigned toothpaste and were instructed to follow the same brushing protocol for the entire month as well as a brushing diary to assist in recording daily participation.

The identical procedures were repeated at the 30 day follow up visit.. In addition, the Plaque HD group was instructed to brush in front of a mirror for 1 minute and to concentrate on removing all visible dye. The placebo group was asked to brush their teeth for 1 minute in front of a mirror, using the provided manual toothbrush.

.

ELIGIBILITY:
Inclusion Criteria:

The inclusion criteria were as follows:

* Apparently healthy men and women age 19-45 with no history of CVD
* All 12 anterior teeth present (canine to canine in both upper and lower arches)
* English speaking
* Ability to commit to two 30 minute appointments These appointment must be 1 month apart)

Exclusion Criteria:

* • Student, faculty or staff with a clinical role at the University of Illinois College of Dentistry
* Individuals taking aspirin, other non-steroidal anti-inflammatory drugs or statins.
* Women who are pregnant or nursing
* Women taking birth control pills or using any hormone released birth control device
* Women on hormone replacement therapy
* Individuals who have taken antibiotics within two weeks of data collection appointment
* Individuals experiencing xerostomia
* Individuals who have experienced an illness, infection or tissue injury within two weeks of data collection appointment
* Individuals with arthritis, lupus or other chronic inflammatory conditions or syndromes
* Individuals with allergies to dyes or over the counter products
* Individuals who have missing anterior teeth, fixed or removable appliances or visible decay or staining in the anterior region (canine to canine in both upper and lower arches)
* Individuals whom have had a dental prophylaxis within 30 days of the data collection visit
* Individuals who have had a new restoration placed (anywhere in the oral cavity) within 30 days of the data collection visit

Ages: 19 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 61 (Actual)
Dates: Start 2015-09-01 (Actual); Primary Completion 2016-04-01 (Actual); Study Completion 2016-08-22 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Kimberly Fasula, MS, Principal Investigator — University of Illinois at Chicago
Locations (1):
- UIC Clinical Research Center, Chicago, Illinois, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Kim YH, Lee SY. Identification of non-streptococcal organisms from human dental plaque grown on the Streptococcus-selective medium mitis-salivarius agar. Arch Oral Biol. 2015 Feb;60(2):267-71. doi: 10.1016/j.archoralbio.2014.11.002. Epub 2014 Nov 8. PMID 25463904
- [Background] de Oliveira C, Watt R, Hamer M. Toothbrushing, inflammation, and risk of cardiovascular disease: results from Scottish Health Survey. BMJ. 2010 May 27;340:c2451. doi: 10.1136/bmj.c2451. PMID 20508025
- [Background] Kholy KE, Genco RJ, Van Dyke TE. Oral infections and cardiovascular disease. Trends Endocrinol Metab. 2015 Jun;26(6):315-21. doi: 10.1016/j.tem.2015.03.001. Epub 2015 Apr 16. PMID 25892452
- [Background] Mbawalla HS, Masalu JR, Astrom AN. Socio-demographic and behavioural correlates of oral hygiene status and oral health related quality of life, the Limpopo-Arusha school health project (LASH): a cross-sectional study. BMC Pediatr. 2010 Nov 30;10:87. doi: 10.1186/1471-2431-10-87. PMID 21118499
- [Background] Gundala R, Chava VK. Effect of lifestyle, education and socioeconomic status on periodontal health. Contemp Clin Dent. 2010 Jan;1(1):23-6. doi: 10.4103/0976-237X.62516. PMID 22114373
- [Background] Al-Anezi SA, Harradine NW. Quantifying plaque during orthodontic treatment: Angle Orthod. 2012 Jul;82(4):748-53. doi: 10.2319/050111-312.1. Epub 2011 Nov 1. PMID 22044115
- [Background] Carter K, Landini G, Walmsley AD. Automated quantification of dental plaque accumulation using digital imaging. J Dent. 2004 Nov;32(8):623-8. doi: 10.1016/j.jdent.2004.06.006. PMID 15476956
- [Background] Short VL, Ivory-Walls T, Smith L, Loustalot F. The Mississippi Delta Cardiovascular Health Examination Survey: Study Design and Methods. Epidemiol Res Int. 2014 Jan 1;2014(Article 499 861461):861461. doi: 10.1155/2014/861461. PMID 25844257
- [Background] Mozaffarian D, Benjamin EJ, Go AS, Arnett DK, Blaha MJ, Cushman M, de Ferranti S, Despres JP, Fullerton HJ, Howard VJ, Huffman MD, Judd SE, Kissela BM, Lackland DT, Lichtman JH, Lisabeth LD, Liu S, Mackey RH, Matchar DB, McGuire DK, Mohler ER 3rd, Moy CS, Muntner P, Mussolino ME, Nasir K, Neumar RW, Nichol G, Palaniappan L, Pandey DK, Reeves MJ, Rodriguez CJ, Sorlie PD, Stein J, Towfighi A, Turan TN, Virani SS, Willey JZ, Woo D, Yeh RW, Turner MB; American Heart Association Statistics Committee and Stroke Statistics Subcommittee. Heart disease and stroke statistics--2015 update: a report from the American Heart Association. Circulation. 2015 Jan 27;131(4):e29-322. doi: 10.1161/CIR.0000000000000152. Epub 2014 Dec 17. No abstract available. PMID 25520374
- [Background] Anderson KM, Odell PM, Wilson PW, Kannel WB. Cardiovascular disease risk profiles. Am Heart J. 1991 Jan;121(1 Pt 2):293-8. doi: 10.1016/0002-8703(91)90861-b. PMID 1985385
- [Background] Loos BG, Craandijk J, Hoek FJ, Wertheim-van Dillen PM, van der Velden U. Elevation of systemic markers related to cardiovascular diseases in the peripheral blood of periodontitis patients. J Periodontol. 2000 Oct;71(10):1528-34. doi: 10.1902/jop.2000.71.10.1528. PMID 11063384
- [Background] Danesh J, Wheeler JG, Hirschfield GM, Eda S, Eiriksdottir G, Rumley A, Lowe GD, Pepys MB, Gudnason V. C-reactive protein and other circulating markers of inflammation in the prediction of coronary heart disease. N Engl J Med. 2004 Apr 1;350(14):1387-97. doi: 10.1056/NEJMoa032804. PMID 15070788
- [Background] Ramamoorthy RD, Nallasamy V, Reddy R, Esther N, Maruthappan Y. A review of C-reactive protein: A diagnostic indicator in periodontal medicine. J Pharm Bioallied Sci. 2012 Aug;4(Suppl 2):S422-6. doi: 10.4103/0975-7406.100318. PMID 23066303
- [Background] D'Aiuto F, Parkar M, Andreou G, Suvan J, Brett PM, Ready D, Tonetti MS. Periodontitis and systemic inflammation: control of the local infection is associated with a reduction in serum inflammatory markers. J Dent Res. 2004 Feb;83(2):156-60. doi: 10.1177/154405910408300214. PMID 14742655
- [Background] Noack B, Genco RJ, Trevisan M, Grossi S, Zambon JJ, De Nardin E. Periodontal infections contribute to elevated systemic C-reactive protein level. J Periodontol. 2001 Sep;72(9):1221-7. doi: 10.1902/jop.2000.72.9.1221. PMID 11577954
- [Background] Ridker PM, Hennekens CH, Buring JE, Rifai N. C-reactive protein and other markers of inflammation in the prediction of cardiovascular disease in women. N Engl J Med. 2000 Mar 23;342(12):836-43. doi: 10.1056/NEJM200003233421202. PMID 10733371
- [Background] Ridker PM, Cushman M, Stampfer MJ, Tracy RP, Hennekens CH. Inflammation, aspirin, and the risk of cardiovascular disease in apparently healthy men. N Engl J Med. 1997 Apr 3;336(14):973-9. doi: 10.1056/NEJM199704033361401. PMID 9077376
- [Background] Pepys MB, Hirschfield GM. C-reactive protein: a critical update. J Clin Invest. 2003 Jun;111(12):1805-12. doi: 10.1172/JCI18921. No abstract available. PMID 12813013
- [Background] Van Dyke TE, van Winkelhoff AJ. Infection and inflammatory mechanisms. J Clin Periodontol. 2013 Apr;40 Suppl 14:S1-7. doi: 10.1111/jcpe.12088. PMID 23627321
- [Background] Kim HC, Yang DM, Lee CM, Jin W, Nam DH, Song JY, Kim JY. Acute appendicitis: relationships between CT-determined severities and serum white blood cell counts and C-reactive protein levels. Br J Radiol. 2011 Dec;84(1008):1115-20. doi: 10.1259/bjr/47699219. Epub 2010 Dec 1. PMID 21123307
- [Background] Pejcic A, Kesic LJ, Milasin J. C-reactive protein as a systemic marker of inflammation in periodontitis. Eur J Clin Microbiol Infect Dis. 2011 Mar;30(3):407-14. doi: 10.1007/s10096-010-1101-1. Epub 2010 Nov 6. PMID 21057970
- [Background] Cusumano CA. Periodontal disease associated with an increased CRP in chronic hemodialysis patients. Rev Nefrol Dial Trans. 2013; 33:188-195.
- [Background] Loos BG. Systemic markers of inflammation in periodontitis. J Periodontol. 2005 Nov;76(11 Suppl):2106-15. doi: 10.1902/jop.2005.76.11-S.2106. PMID 16277583
- [Background] Tonetti MS. Periodontitis and risk for atherosclerosis: an update on intervention trials. J Clin Periodontol. 2009 Jul;36 Suppl 10:15-9. doi: 10.1111/j.1600-051X.2009.01417.x. PMID 19432627
- [Background] Persson GR, Persson RE. Cardiovascular disease and periodontitis: an update on the associations and risk. J Clin Periodontol. 2008 Sep;35(8 Suppl):362-79. doi: 10.1111/j.1600-051X.2008.01281.x. PMID 18724863
- [Background] Goyal L, Bey A, Gupta ND, Sharma VK. Comparative evaluation of serum C-reactive protein levels in chronic and aggressive periodontitis patients and association with periodontal disease severity. Contemp Clin Dent. 2014 Oct;5(4):484-8. doi: 10.4103/0976-237X.142816. PMID 25395764
- [Background] Kumar KR, Ranganath V, Naik R, Banu S, Nichani AS. Assessment of high-sensitivity C-reactive protein and lipid levels in healthy adults and patients with coronary artery disease, with and without periodontitis--a cross-sectional study. J Periodontal Res. 2014 Dec;49(6):836-44. doi: 10.1111/jre.12172. Epub 2014 Mar 12. PMID 24620793
- [Background] Anitha G, Nagaraj M, Jayashree A. Comparative evaluation of levels of C-reactive protein and PMN in periodontitis patients related to cardiovascular disease. J Indian Soc Periodontol. 2013 May;17(3):330-2. doi: 10.4103/0972-124X.115657. PMID 24049333
- [Background] Zijnge V, van Leeuwen MB, Degener JE, Abbas F, Thurnheer T, Gmur R, Harmsen HJ. Oral biofilm architecture on natural teeth. PLoS One. 2010 Feb 24;5(2):e9321. doi: 10.1371/journal.pone.0009321. PMID 20195365
- [Background] Chen T, Yu WH, Izard J, Baranova OV, Lakshmanan A, Dewhirst FE. The Human Oral Microbiome Database: a web accessible resource for investigating oral microbe taxonomic and genomic information. Database (Oxford). 2010 Jul 6;2010:baq013. doi: 10.1093/database/baq013. PMID 20624719
- [Background] Bokhari SA, Khan AA, Butt AK, Azhar M, Hanif M, Izhar M, Tatakis DN. Non-surgical periodontal therapy reduces coronary heart disease risk markers: a randomized controlled trial. J Clin Periodontol. 2012 Nov;39(11):1065-74. doi: 10.1111/j.1600-051X.2012.01942.x. Epub 2012 Sep 11. PMID 22966824
- [Background] Kajikawa M, Nakashima A, Maruhashi T, Iwamoto Y, Iwamoto A, Matsumoto T, Hidaka T, Kihara Y, Chayama K, Goto C, Taguchi A, Noma K, Higashi Y. Poor oral health, that is, decreased frequency of tooth brushing, is associated with endothelial dysfunction. Circ J. 2014;78(4):950-4. doi: 10.1253/circj.cj-13-1330. Epub 2014 Feb 5. PMID 24500034
- [Background] Mani A, Vadvadgi V, Anarthe R, Saini R, Mani S. A clinical study on Dental Air Force Cleaning System on adult chronic periodontits and its assessment to C-reactive protein levels. Int J Exp Dent Sci. 2012; 1:14-18.
- [Background] Harnacke D, Winterfeld T, Erhardt J, Schlueter N, Ganss C, Margraf-Stiksrud J, Deinzer R. What is the best predictor for oral cleanliness after brushing? Results from an observational cohort study. J Periodontol. 2015 Jan;86(1):101-7. doi: 10.1902/jop.2014.140152. PMID 25186778
- [Background] Stevens K, Belavsky B, Evans CA, Viana MG, Wu C. Evaluation of plaque removal efficacy of a novel dye-containing toothpaste: a clinical trial. Int J Dentistry Oral Sci. 2016; 3(1):185-189
- See also: The World Health Organization. Cardiovascular Diseases (CVDs) — http://www.who.int/cardiovascular_diseases/en/
- See also: American Heart Association. Heart and Stroke Statistics. — http://www.heart.org/HEARTORG/General/Heart-and-Stroke-Association-Statistics_UCM_319064_SubHomePage.jsp.
- See also: Relationship between serum antibody titres to porphyromonas gingivalis and hs-CRP levels as inflammatory markers of periodontitis. — http://www.sciencedirect.com.proxy.cc.uic.edu/science/article/pii/S0003996911003876
- See also: HSRIC: Grants, funding and fellowships. — http://www.nlm.nih.gov/hsrinfo/grantsites.html

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Sixty-one apparently healthy subjects aged 19-45 were recruited from the University of Illinois at Chicago campus and surrounding Medical District. Recruitment began in August 2015.
Pre-assignment Details: This study did not include pre-assignment criteria other than inclusion/exclusion criteria that determined study eligibility. Only 5 of the 66 screened subjects did not meet eligibility for participation. Qualified subjects were then assigned, by computer randomization in Crosspad©, a subject identification number and randomized.
Groups:
- Plaque Identifying Toothpaste: A 30 day supply of dosed syringes containing a plaque identifying toothpaste. Toothpaste was dosed in 2 ml syringes and subjects were instructed to use half (1ml) in the morning and half (1ml) in the evening.
- Non-plaque Identifying Toothpaste: A 30 day supply of dosed syringes containing an identical non-plaque identifying toothpaste. Toothpaste was dosed in 2 ml syringes and subjects were instructed to use half (1ml) in the morning and half (1ml) in the evening.
Period: Overall Study
Arm/Group | Plaque Identifying Toothpaste | Non-plaque Identifying Toothpaste
Started | 31 | 30
Completed | 31 | 30
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: Baseline plaque score was assessed using DPIA and baseline inflammation was assessed using hs-CRP
Groups:
- Plaque Identifying Toothpaste: A 30 day supply of dosed syringes containing a plaque identifying toothpaste
  Plaque identifying toothpaste: Plaque identifying toothpaste
  Toothpaste is dosed in 2 ml syringes and subjects were instructed to use half (1ml) in the morning and half (1ml) in the evening.
- Non-plaque Identifying Toothpaste: A 30 day supply of dosed syringes containing an identical non-plaque identifying toothpaste
  Non-plaque identifying toothpaste: Non-plaque identifying toothpaste
  Toothpaste is dosed in 2 ml syringes and subjects were instructed to use half (1ml) in the morning and half (1ml) in the evening.
- Total: Total of all reporting groups
Arm/Group | Plaque Identifying Toothpaste | Non-plaque Identifying Toothpaste | Total
Number analyzed (Participants) | 31 | 30 | 61
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 31 | 30 | 61
  >=65 years | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 16 | 18 | 34
  Male | 15 | 12 | 27
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Race/Ethnicity: African American | 6 | 5 | 11
  Race/Ethnicity: Asian | 13 | 10 | 23
  Race/Ethnicity: Caucasian | 8 | 8 | 16
  Race/Ethnicity: Hispanic | 4 | 7 | 11
  Race/Ethnicity: Other | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 31 | 30 | 61
Digital Plaque Image Analysis (DPIA) [Geometric Mean (Standard Deviation); unit: log(Percentage)] — log(100% * (plaque pixels) / (plaque + teeth pixels))
  log(Percentage) | 1.69 (1.21) | 1.06 (1.58) | 1.38 (1.43)
High-sensitivity C-Reactive Protein (hs-CRP) [Geometric Mean (Standard Deviation); unit: log(mg/L)] | 0.10 (1.30) | 0.24 (1.17) | 0.17 (1.23)

OUTCOME MEASURES:

1. Primary Outcome: Change in Oral Plaque
Description: Measure description "percentage" refers to the change in plaque percentage from the baseline to the follow-up visit. The follow-up visit occurred between 30 and 60 days post baseline.
Time Frame: Baseline to 30 - 60 days post baseline
Population: Primary analysis group definition was based on the Intent-to-Treat (ITT) principle.
Measure: Geometric Mean (95% Confidence Interval); unit: log(percentage)
Arm/Group | Plaque Identifying Toothpaste | Non-plaque Identifying Toothpaste
Number analyzed (Participants) | 31 | 30
log(percentage) | -1.05 [-1.45 to -0.66] | -0.03 [-0.43 to 0.38]
Statistical Analysis 1: Comparison: Plaque Identifying Toothpaste vs Non-plaque Identifying Toothpaste; Test type: Other — Test conducted was a test of difference between plaque identifying toothpaste and non-plaque identifying toothpaste for change in DPIA from pre to post; p = 0.001, Repeated Measures ANOVA; Mean Difference (Net) = -1.02, 95% CI 2-sided [-1.60 to -0.44]

2. Primary Outcome: Change in Hs-CRP Serum Level
Description: Measure description "mg/L" refers to the change in hs-CRP per mg/L from the baseline to the follow-up visit. The follow-up visit occurred between 30 and 60 days post baseline.
Time Frame: Baseline to 30 - 60 days post baseline
Population: Primary analysis group definition was based on the Intent-to-Treat (ITT) principle.
Measure: Geometric Mean (95% Confidence Interval); unit: log(mg/L)
Arm/Group | Plaque Identifying Toothpaste | Non-plaque Identifying Toothpaste
Number analyzed (Participants) | 31 | 30
log(mg/L) | 0.04 [-0.31 to 0.38] | 0.22 [-0.13 to 0.58]
Statistical Analysis 1: Comparison: Plaque Identifying Toothpaste vs Non-plaque Identifying Toothpaste; Test type: Other — Test conducted was a test of the difference between plaque identifying toothpaste and non-plaque identifying toothpaste for change in hsCRP; p = 0.459, Repeated Measures ANOVA; Mean Difference (Net) = -0.18, 95% CI 2-sided [-0.69 to 0.32]

3. Secondary Outcome: Change in Oral Plaque - PSS Analysis
Description: Measure description "percentage" refers to the change in plaque percentage from the baseline to the follow-up visit. The follow-up visit occurred between 30 and 60 days post baseline for the Pre-Specified Subgroup (PSS).
Time Frame: Baseline to 30-60 days post
Population: Secondary analysis group definition was based on Pre-Specified Subgroup of subjects such that 30 <= follow-up <= 60 days
Measure: Geometric Mean (95% Confidence Interval); unit: log(percentage)
Groups:
- Plaque Identifying Toothpaste: A 30 day supply of daily syringes containing a plaque identifying toothpaste with targetol
  Plaque identifying toothpaste: Plaque identifying toothpaste with targetol
  With follow-up between 30-60 days.
- Non-plaque Identifying Toothpaste: A 30 day supply of daily syringes containing an identical non plaque identifying toothpaste without targetol
  Non-plaque identifying toothpaste: Non-plaque identifying toothpaste without targetol
  With follow-up between 30-60 days.
Arm/Group | Plaque Identifying Toothpaste | Non-plaque Identifying Toothpaste
Number analyzed (Participants) | 31 | 29
log(percentage) | -1.05 [-1.44 to -0.66] | -0.10 [-0.50 to 0.31]

4. Secondary Outcome: Change in Inflammation - PSS Analysis
Description: Measure description "mg/L" refers to the change in hs-CRP per mg/L from the baseline to the follow-up visit. The follow-up visit occurred between 30 and 60 days post baseline. -PSS analysis
Time Frame: Baseline to 30-60 days post
Population: Secondary analysis group definition for hs-CRP was based on a Pre-Specified Subgroup which had 0.5 <= baseline hs-CRP <= 10.0 and 30 <= follow-up <= 60 days
Measure: Geometric Mean (95% Confidence Interval); unit: log(mg/L)
Groups:
- Plaque Identifying Toothpaste: A 30 day supply of daily syringes containing a plaque identifying toothpaste with targetol
  Plaque identifying toothpaste: Plaque identifying toothpaste with targetol
  With baseline hs-CRP between 0.5 and 10 mg/L and follow-up between 30-60 days.
- Non-plaque Identifying Toothpaste: A 30 day supply of daily syringes containing an identical non plaque identifying toothpaste without targetol
  Non-plaque identifying toothpaste: Non-plaque identifying toothpaste without targetol
  With baseline hs-CRP between 0.5 and 10 mg/L and follow-up between 30-60 days.
Arm/Group | Plaque Identifying Toothpaste | Non-plaque Identifying Toothpaste
Number analyzed (Participants) | 19 | 19
log(mg/L) | -0.40 [-0.75 to -0.04] | 0.14 [-0.21 to 0.50]

ADVERSE EVENTS:
Time Frame: Baseline to follow-up (30 - 60 days post baseline)
Description: Adverse events were identified as:
  1. All-Cause Mortality
  2. Serious Adverse Events
  3. Other (Not Including Serious) Adverse Events
  Subjects were instructed to discontinue toothpaste use and contact PI if they experienced any adverse reactions to the product. Subjects were instructed to call 911 if any serious reactions occurred. Subjects were asked at follow-up visit and post-study debriefing if any adverse events occurred.
  No adverse events were reported.
Groups:
- Plaque Identifying Toothpaste: A 30 day supply of dosed syringes containing a plaque identifying toothpaste
  Plaque identifying toothpaste: Plaque identifying toothpaste
- Non-plaque Identifying Toothpaste: A 30 day supply of dosed syringes containing an identical non plaque identifying toothpaste
  Non-plaque identifying toothpaste: Non-plaque identifying toothpaste
Arm/Group | Plaque Identifying Toothpaste | Non-plaque Identifying Toothpaste
All-Cause Mortality (participants affected / at risk) | 0/31 | 0/30
Serious Adverse Events (participants affected / at risk) | 0/31 | 0/30
Other Adverse Events (participants affected / at risk) | 0/31 | 0/30

LIMITATIONS AND CAVEATS:
Funding limited the study to a small number of subjects. Funding also limited options to compensate subject as a method to pre-select subjects with elevated hs-CRP.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No